CLINICAL TRIAL: NCT01016522
Title: Safety and Tolerability of the Ketogenic Diet in ALS
Brief Title: Safety and Tolerability of the Ketogenic Diet in Amyotrophic Lateral Sclerosis (ALS)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Nutricia North America (Industry); Cornell University (Other)
Responsible Party: Principal Investigator, Vinay Chaudhry, Professor, Johns Hopkins University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NA_00008855; NCT01035710 (obsolete NCT alias)
Record Dates: First submitted 2009-11-18; First posted 2009-11-19 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2015-03

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: ALS; Ketogenic Diet
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- KetoCal (Experimental): KetoCal tube feeding formula
  Interventions: Dietary Supplement: KetoCal

INTERVENTIONS:
Dietary Supplement: KetoCal — Ketogenic Diet food via gastrostomy tube - 80% fat, 17% protein, 3% carbohydrates

SUMMARY:
This research is being done to see if the ketogenic diet (which is high in fat and low in carbohydrates) is safe and tolerable in amyotrophic lateral sclerosis (ALS) patients who are fed through a gastrostomy tube. This is not a study to see if ketogenic diets are effective in the treatment of ALS.

ELIGIBILITY:
Inclusion Criteria:

1. Familial or sporadic ALS diagnosed as probable, laboratory-supported probable or definite according to the World Federation of Neurology El Escorial criteria
2. Age 18 or older
3. Capable of providing informed consent and complying with trial procedures
4. Gastrostomy tube in place for the prior month
5. Appel ALS score less than 100
6. Able to stand on a scale with assistance
7. For patients with Appel ALS scores greater than 80, availability of caregiver who is willing and able to:

   * Prepare, administer and log tube feeds
   * Check and log gastric residuals
   * Assist with weighing subject at home if necessary
8. Willing to chart food intake during the six-month study
9. Patients either not taking Riluzole (Rilutek) or Minocycline or on a stable dose of these for 30 days
10. Not taking Coenzyme Q10 or on a stable dose and brand for 30 days
11. Absence of exclusion criteria

Exclusion Criteria:

1. Forced vital capacity <50% of predicted
2. Dependence on mechanical ventilation for more than 12 hours per day
3. Exposure to any experimental agent within 30 days of onset of this protocol
4. Women who are pregnant or planning to become pregnant
5. Women of childbearing potential not practicing contraception
6. Enrollment in another research study within 30 days of or during this trial
7. Mini-Mental State Exam (MMSE) score <20
8. Patients with symptomatic cardiac disease or hypercholesterolemia
9. Patients with myocardial infarction within 6 months of this trial
10. Renal dysfunction defined as BUN and creatinine >2XULN
11. Known mitochondrial disease
12. BMI<18.5
13. Prior use of a 4:1 ketogenic diet or Atkins diet within 1 month of this trial
14. Impaired liver function, defined as AST or ALT of 3 X ULN
15. Patients who have a pacemaker or other internal electronic medical device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2009-11; Primary Completion 2011-02 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Study will determine if humans with ALS fed a strictly controlled diet designed to generate large amounts of ketones is safe and well-tolerated without evidence of weight loss or other adverse effect | 28 weeks

SECONDARY OUTCOMES:
Evaluate changes in motor function, strength, fatigue, body fat and cognitive function | 28 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Johns Hopkins ALS Clinic, Baltimore, Maryland, United States